CLINICAL TRIAL: NCT04681235
Title: Virtual Reality Training Affects on Motor Functions and Mental Health in Stroke Patients: a Pilot Study
Brief Title: Virtual Reality Training Affects on Motor Functions and Mental Health in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VR001
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Stroke; Motor Disorders; Affective Symptoms; Gait Disorder, Sensorimotor
Keywords: Stroke; Virtual reality; Rehabilitation; Motion capture
MeSH Terms: conditions — Stroke; Motor Disorders; Affective Symptoms; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Group (Experimental): Training Group recieved 10 sessions on VR (Grail Motekforce, Netherlands) during two weeks. One session lasted 40 minuties.
  Interventions: Other: Training on VR

INTERVENTIONS:
Other: Training on VR — The training is aimed at improving the functioning of the motor sphere, including balance, gait, and upper limb function, as well as increasing the level of motivation and reducing the level of anxiety and depression. Game applications were selected based on therapeutic tasks of motor recovery.

SUMMARY:
In our study, we tested the hypothesis of the safe effect applicability of motor training in the immersion high-tech polymodal VR system not only on the parameters of balance, gait, and motor status of the patient, but also on his cognitive functions and mental health in patients with a degree of disability no more than 3 points on a scale Rankin.

DETAILED DESCRIPTION:
The neurological consequences of stroke cover the motor, sensory, visual, affective, cognitive and speech spheres. 55-75% of stroke survivors suffer from motor impairments, caused, inter alia, by hemiparesis, which substantially reduce the quality of their life. In addition, neurocognitive functions, especially memory, visual-constructive abilities and executive functions, are often affected by stroke. Cognitive impairments appear in 83% patients in at least one cognitive domain, whereas in 50% patients appear in multiple (≥3) domains. These disorders affect the quality of life of patients, their skills of daily activity (the ability to go to the store, prepare food, plan their actions for organizing a daily routine), social adaptation. One of the rehabilitation methods that are comprehensively suitable for the recovering on of stroke consequences is the intervention using virtual reality. The VR method is used for the rehabilitation of stroke patients with various motor and neurocognitive deficits: one-sided spatial ignorance, disorders of attention, memory, mood, visual-spatial functions, and constructive abilities.

In our study, we tested the hypothesis of the applicability of the safe effect of motor training in the immersion high-tech polymodal VR system not only on the parameters of balance, gait, and motor status of the patient, but also on his cognitive functions and mental health in patients with a degree of disability no more than 3 score on a modified Rankin Scale.

Stroke patients participated in the study in Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health in Moscow, Russia. The study was run between October 2019 and July 2020 and was approved by a local ethic committee and followed principles of the Declaration of Helsinki. The patients stayed in a 24-hour hospital and underwent a rehabilitation course. This course included a VR Trainig of 10 sessions of 40 minutes each, which the patients took over two weeks. VR training was conducted on the GRAIL system equipment (Motekforce, Netherlands), consisting of a semi-cylindrical screen, treadmill, 10 infrared cameras (Vicon, UK) and reflective markers, and software providing biofeedback in real time. For complex recovery in VR, exercises stimulate the motor, cognitive and behavioral spheres, including visual-spatial orientation, the process of attention (with one and duai-task), executive functions, lowering the level of anxiety, hand-eye coordination and balance.Training applications were based on the therapeutic goals for every patient, according to postural stability and gait adaptation.

Before and after the end of the training, the patient's condition was assessed, including measurements in motor and daily living activity, measurements in mental health, measurements in Virtual Reality.

ELIGIBILITY:
Inclusion Criteria:

with a stroke, transferred at least 2 weeks ago; with no history of neurological or psychiatric disorders; able to maintain an upright posture and walk without support or with minimal support for at least 30 minutes; with stable hemodynamics;

Exclusion Criteria:

not having epileptic activity; not having serious ophthalmic disorders; less than 24 scores in MoCA

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Postural stability test (Grail Motekforce) | Change from baseline at 2 weeks
  The subject's ability to remain balanced under four different conditions is evaluated (cm/s).
Six-minute walk test (6MWT) (Grail Motekforce) | Change from baseline at 2 weeks
  The 6-minute walk test evaluates how much distance a subject can cover in six minutes (m).
Beck Depression Inventory | Change from baseline at 2 weeks
  Measures the severity of depression (0-63; 30-63 scores indicate severe depression)
State-Trait Anxiety Inventory | Change from baseline at 2 weeks
  Examines two types of anxiety - state anxiety (anxiety about an event) and trait anxiety (anxiety level as a personal characteristic) with the score range from 20 to 80, where higher scores correspond to greater anxiety

SECONDARY OUTCOMES:
Standing Balance Test | Change from baseline at 2 weeks
  Examines the patient's ability to maintain an upright position (0-4, where 0 - can't stand)
Berg Balance Scale | Change from baseline at 2 weeks
  Relates to evaluation of static and dynamic balance, consists of 14 tasks, ranging from standing up from a sitting position, to standing on one foot
Timed Up and Go Test | Change from baseline at 2 weeks
  Examines functional mobility and requires a patient to stand up, walk 3 meters, turn, walk back, and sit down; result is obtained in seconds
Hauser Ambulation Index | Change from baseline at 2 weeks
  Assess mobility by evaluating the time and degree of assistance required to walk a 8-m distance as quickly and safely as possible, with scores that range from 0 (asymptomatic) to 10 (bedridden)
Rivermead Activities of Daily Living Scales | Change from baseline at 2 weeks
  Assesses self-service and two types of domestic activities, maximum scores (90) indicate independence in daily living activity
Functional Independence Measure | Change from baseline at 2 weeks
  Examines the functional status of the patient in 18 domains related to cognitive and motor functions up to the maximum in 126 scores (independence in daily life)

CONTACTS AND LOCATIONS:
Overall Officials: Marina A Shurupova, Principal Investigator — Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health; Alina D Aizenshtein, Principal Investigator — Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health; Galina Ivanova, Prof., Study Chair — Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health; Nadezhda L Cherepahina, PhD, Principal Investigator — Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health
Locations (1):
- Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No